CLINICAL TRIAL: NCT00929357
Title: A Retrospective Evaluation of the Radiographic Efficacy of Different Conventional Systemic Therapies and Biologics in Patients With Rheumatoid Arthritis in Routine Practice.
Brief Title: Retrospective Evaluation of the Radiographic Efficacy of Conventional and Biologic Treatment
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Wyeth
Other Study IDs: 0881X1-4617
Record Dates: First submitted 2009-06-25; First posted 2009-06-29 (Estimated); Results first posted 2011-06-28 (Estimated); Last update posted 2011-08-10 (Estimated); Status verified 2011-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Antirheumatic Agents; Biological Products

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- 1: DMARDs
  Interventions: Drug: DMARDs or Biologics
- 2: Biologics
  Interventions: Drug: DMARDs or Biologics

INTERVENTIONS:
Drug: DMARDs or Biologics

SUMMARY:
This study involves review and analysis of disease activity in patients with rheumatoid arthritis who where treated with either conventional DMARDs (Disease Modifying Antirheumatic Drugs) or Biologics and have two existing, consecutive radiographs (x-ray images) of hand and feet taken as part of routine treatment monitoring within a time interval of 12 to 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Secure diagnosis of rheumatoid arthritis
* Older than 18 years
* Two consecutive plain radiographs of the hands and feet with a time interval of 12 to 36 months are available. The radiographs are recorded 2003 or later and are in accordance with a defined X-ray protocol.

Exclusion Criteria:

- Patients who receive Anakinra, Rituximab or Abatacept

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 200
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2009-08; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Schmittingheide 20-32, Munster, Denmark

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 160 participants were screened and 156 entered this non-randomized retrospective evaluation of conventional systemic therapies and biologics in participants with rheumatoid arthritis in routine practice.
Pre-assignment Details: Participants had been treated according to authorized dosages for disease-modifying anti-rheumatic drug (DMARDs) and biologics in Germany. No investigational product had been provided.
Groups:
- DMARDS: Participants had received disease-modifying basic Rheumatoid Arthritis (RA) therapy with a conventional anti-rheumatic drug (DMARDS) such as methotrexate, leflunomide, or a combination of these.
- Biologics: Participants had received disease-modifying basic Rheumatoid Arthritis (RA) therapy with a tumor necrosis factor (TNF)-alpha-blocker such as etanercept (Enbrel®), infliximab (Remicade®) or adalimumab (Humira®) - may be administered in combination with a conventional DMARD.
Period: Overall Study
Arm/Group | DMARDS | Biologics
Started | 92 | 64
Completed | 92 | 64
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DMARDS | Biologics | Total
Number analyzed (Participants) | 92 | 64 | 156
Age, Customized [Mean (Standard Deviation); unit: years] | 61.6 (12.6) | 58.9 (13.1) | 60.5 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 50 | 113
  Male | 29 | 14 | 43

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Joint Status Assessed by Radiographic (Roentgen) Progression
Description: Radiographic progression assessed using Ratingen score with range of 0 = normal joint; 1 = one or more erosions, <20% of the joint surface are destroyed; 2 = 21% to 40% of the joint surface are destroyed; 3 = 41% to 60% of joint surface are destroyed; 4 = 61% to 80% of the joint surface are destroyed; 5 = >80% of the joint surface are destroyed. Total possible score based on 38 joints was 0 to 190; higher scores indicated greater joint destruction. Annualized change in Ratingen score calculated as (total change in Ratingen score / time period between radiograph 1 and 2 [months])*12 months.
Time Frame: Baseline (Day 0) up to 48 months
Population: Evaluable population: all participants who had provided two evaluable, consecutive radiographs of the hands and forefeet, taken at intervals of 12 to 48 months. Since the time period between the first and second radiograph could range between 12 to 48 months, changes in Ratingen score were to be normalized to 1 year.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | DMARDS | Biologics
Number analyzed (Participants) | 92 | 64
scores on a scale
  Baseline Ratingen score - first radiograph | 6.9 (10.7) | 24.3 (30.7)
  Change at second radiograph | 0.0 (3.0) | 0.3 (6.3)
  Annualized change in Ratingen score | -0.1 (1.4) | 0.0 (3.3)

2. Secondary Outcome: Number of Participants Without Radiographic Progression
Description: An increase of 4 or more points in the Ratingen score was necessary to detect a difference in radiographic progression. Ratingen score range 0 = normal joint to 5 = >80% of the joint surface are destroyed. Total possible score based on 38 joints was 0 to 190; higher scores indicated greater joint destruction. A decrease of 4 (smallest detectable difference) or more points in total Ratingen score was considered a decrease in erosive damage.
Time Frame: Baseline (Day 0) up to 48 months
Population: Evaluable population
Measure: Number; unit: participants
Arm/Group | DMARDS | Biologics
Number analyzed (Participants) | 92 | 64
participants | 89 | 59

3. Secondary Outcome: Number of Participants Without Erosions
Description: Radiographic assessment of no erosions using Ratingen scoring categorized as score of 0=normal joint.
Time Frame: Baseline (Day 0) up to 48 months
Population: Evaluable population. Ratingen scores were calculated based on radiographic assessment, but score of 0 (no erosions) was not reported separately; data not summarized.
Measure: Number; unit: participants
Arm/Group | DMARDS | Biologics
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change From Baseline in Disease Activity Score Based on 28 Joints (DAS 28)
Description: DAS28 calculated from the number of swollen joints (SJC) and painful joints (PJC) using the 28 joints count, the erythrocyte sedimentation rate (ESR) (millimeters per hour [mm/hour]) and patient's global assessment (PGA) of disease activity (participant rated arthritis activity assessment with transformed scores ranging 0 to 10; higher scores indicated greater affectation due to disease activity). DAS28 ≤3.2 = low disease activity, DAS28 >3.2 to 5.1 = moderate to high disease activity.
Time Frame: Baseline (Day 0) up to 48 months
Population: Evaluable population; (n)=number of participants with analyzable data at observation for DMARDS and Biologics, respectively.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | DMARDS | Biologics
Number analyzed (Participants) | 92 | 64
scores on a scale
  Baseline DAS 28 - first radiograph (n=85, 61) | 4.0 (1.7) | 4.0 (1.7)
  Change at second radiograph (n=83, 58) | -0.8 (1.6) | -0.7 (1.5)

5. Secondary Outcome: Change From Baseline in Erythrocyte Sedimentation Rate (ESR)
Description: Erythrocyte Sedimentation Rate measured as millimeters per hour (mm/h).
Time Frame: Baseline (Day 0) up to 48 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mm/h
Arm/Group | DMARDS | Biologics
Number analyzed (Participants) | 92 | 64
mm/h
  Baseline ESR - first radiograph (n=91, 63) | 23.8 (21.1) | 22.3 (20.5)
  Change at second radiograph (n=90, 63) | -3.2 (21.8) | 0.3 (19.7)

6. Secondary Outcome: Change From Baseline in C-reactive Protein (CRP)
Description: C-reactive protein measured as milligrams per liter (mg/l)
Time Frame: Baseline (Day 0) up to 48 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg/l
Arm/Group | DMARDS | Biologics
Number analyzed (Participants) | 92 | 64
mg/l
  Baseline CRP- first radiograph (n=90, 64) | 12.9 (20.2) | 12.9 (20.6)
  Change at second radiograph (n=89, 64) | -5.4 (22.6) | -4.3 (21.5)

7. Secondary Outcome: Number of Participants With Change From Baseline in Rheumatoid Factor (RF)
Description: Rheumatoid Factor measured as a titer and categorized as negative (<1:16 ratio) or positive. A ratio >1:16 indicates a higher level of RF.
Time Frame: Baseline (Day 0) up to 48 months
Population: Evaluable population; (n)=number of participants with analyzable data at observation for Positive or Negative status for DMARDS and Biologics, respectively.
Measure: Number; unit: participants
Arm/Group | DMARDS | Biologics
Number analyzed (Participants) | 92 | 64
participants
  Baseline Positive RF- first radiograph (n=89, 62) | 52 | 46
  Baseline Negative RF- first radiograph | 37 | 16
  Positive RF at second radiograph (n=85, 61) | 47 | 49
  Negative RF at second radiograph | 38 | 12

8. Secondary Outcome: Number of Participants With Laboratory Result for Cyclic Citrullinated Peptide-autoantibody-test (CCP)
Description: Cyclic citrullinated peptide-autoantibody-test measured as Enzyme-linked immunosorbent assay (ELISA units or EU) and categorized as negative (<20 EU) or positive (≥20 up to >60 EU).
Time Frame: Baseline (Day 0) up to 48 months
Population: Evaluable population; N=number of participants with evaluable data for CCP. CCP value as a laboratory diagnostic marker was collected within the complete timeframe and was documented only once; calculation for change in value not applicable.
Measure: Number; unit: participants
Arm/Group | DMARDS | Biologics
Number analyzed (Participants) | 85 | 64
participants
  Positive CCP | 50 | 53
  Negative CCP | 35 | 11

ADVERSE EVENTS:
Time Frame: Baseline up to 48 months
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. Event may be categorized as serious in 1 subject and as nonserious in another subject, or 1 subject may have experienced both a serious and nonserious event during the study. No safety evaluation was performed nor intended; no events were reported.
Arm/Group | DMARDS | Biologics
Serious Adverse Events (participants affected / at risk) | 0/92 | 0/65
Other Adverse Events (participants affected / at risk) | 0/92 | 0/65

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.